CLINICAL TRIAL: NCT01462981
Title: Cohort of Hepatitis B Research of Amsterdam
Acronym: COBRA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Public Health Service of Amsterdam (Other Government)
Collaborators: UMC Utrecht (Other)
Responsible Party: Principal Investigator, S. Harkisoen, MD, Public Health Service of Amsterdam
Other Study IDs: COBRA
Record Dates: First submitted 2011-10-28; First posted 2011-11-01 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-11

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Serum, White cells
Oversight: Data Monitoring Committee: No

SUMMARY:
Hepatitis B is a form of liver disease caused by a DNA-virus, called hepatitis B virus (HBV). Infection can result in an inflammation of the liver parenchyma with various clinical manifestations ranging from an asymptomatic course to jaundice. After contact with the virus the immunological response of the host determines the clinical outcome leading to either viral clearance or a chronic infection.

Although several factors are responsible for the development of chronic HBV-infection, one of the factors is a weak and transient CD8+ T-cell responses after HBV infection. In chronic hepatitis B, inflammation can lead to scarring which is the driving force to fibrosis and cirrhosis. Some immunological parameters, like a newly discovered subset of IL-17 producing T helper cells (Th17 cells), may influence the disease progression of HBV. In the cirrhotic patient, eventually there is an increased risk of hepatocellular carcinoma (HCC) leading to liver failure.

Recent literature in Asian patients with chronic hepatitis B showed that serum HBV viral load is a strong predictor for the development of cirrhosis, independent of hepatitis B e- antigen status and serum alanine transaminase level. It is unclear whether these results can be extrapolated to non-Asian (Caucasian and African) populations because of differences in host (HLA background) and viral (HBV genotype) factors.

The aim of this study is to elucidate the question whether historic HBV viral load is associated with the risk of HBV-related cirrhosis or mortality in a cohort of non-Asian individuals with chronic hepatitis B infection.

DETAILED DESCRIPTION:
During one visit, the nurse will assess the quality of life of the included patients with the use of a health assessment questionnaire. This questionnaire is derived from a standardized questionnaire to assess the quality of life in patients, the SF-36. Participation will require a single visit to the outpatient clinic of Public Health Service. During this visit a short history and physical examination related to chronic liver disease will be performed. During the same visit a single venapunction and a single hepatic elastography (fibroscan) will be performed.

ELIGIBILITY:
Inclusion Criteria:

* HBsAg-positivity
* Serum sample available from the screening programme at the Public Health Service
* Still living and alive in Amsterdam or Diemen and address traceable by general practitioners or municipal authorities.
* Non-Asian (both parents not born in Asia)
* Between 18-65 years old
* Capable of giving informed consent and capable of traveling to the Public Health Service

Exclusion Criteria:

* Subjects coinfected with human immunodeficiency virus (HIV)
* Subjects coinfected with hepatitis D virus (HDV)
* Subjects coinfected with hepatitis C virus (HCV)
* Subjects who are unable to come to the outpatient clinic
* Subjects incapable to give informed consent due to legally incompetence

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women between 18 - 65 year in the study period with chronic hepatitis B who were HBsAg positive during pregnancy screening of which serum samples are stored at the Public Health Service.
Sampling Method: Non-Probability Sample
Enrollment: 172 (Estimated)
Dates: Start 2011-09; Study Completion 2012-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Andy IM Hoepelman, MD, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- Public Health Service (GGD), Amsterdam, North Holland, Netherlands